CLINICAL TRIAL: NCT03758053
Title: Stress Sensitivity, Emotion Processing and Cue-reactivity: the Influence of Adverse Childhood Experiences in Substance-related Disorders
Brief Title: Adverse Childhood Experiences in Substance-related Disorders
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: GRK2350-B5
Record Dates: First submitted 2018-08-20; First posted 2018-11-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Alcohol Use Disorder; Trauma, Psychological
MeSH Terms: conditions — Alcoholism; Psychological Trauma | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva (stress hormones) Blood (genotyping)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Individuals with alcohol use disorder + ACE: Individuals with AUD and varying levels of adverse childhood experiences (ACE)
  Interventions: Other: No intervention
- Healthy controls: Healthy individuals without AUD
  Interventions: Other: No intervention
- Individuals with alcohol use disorder, no ACE: Individuals with AUD and no adverse childhood experiences (ACE)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention
  Other Names: observational study

SUMMARY:
Aversive childhood experiences (ACE) and their relation to the development of an alcohol use disorder will be measured with fMRI.

DETAILED DESCRIPTION:
The aim of this study is to examine the impact of ACE on stress sensitivity, cue-reactivity and emotion processing in individuals with AUD. (Neuro-) biological and physiological mechanisms underlying AUD after ACE will be studied.

Neural correlates of stress-sensitivity, emotion processing and alcohol cue-reactivity will be assessed using fMRI. Furthermore, blood and saliva samples will be used to assess biological and physiological mechanisms (e.g. salivary cortisol level or genetic markers of AUD and possible gene-environment-interactions).

The question whether individuals with AUD and ACE might tend to use alcohol to cope with stress, negative affect or intrusions (according to the self-medication model) will be explored. On the other hand, individuals with AUD and low levels of ACE might use alcohol for its positive effects (according to a positive reinforcement model).

90 individuals (30 HC and 60 individuals with AUD and varying levels of ACE) will be examined using interviews, questionnaires and fMRI tasks as well as saliva and blood samples. All ethical votes and informed consents of participants are and will be obtained according to the declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* male and female
* age between 18 and 65
* normal or correctable eyesight
* Sufficient ability to communicate with the investigators, to answer questions in oral and written form
* "Fully Informed Consent"
* "Written Informed Consent"
* Healthy individuals (AUDIT Score<=8, alcohol intake < 12g/ less than 5 days (women) & 24g/ less than 5 days (men)
* Individuals with alcohol use disorder according to DSM-5 or 'heavy drinking' (alcohol intake > 40g/ more than 5 days (women) & 60g/ more than 5 days (men) with up to 28 days of abstinence AND aversive childhood experiences

Exclusion Criteria:

* Withdrawal of the declaration of consent
* Exclusion criteria for an MRI scan (pregnancy, metal implants,...)
* severe internal, neurological and psychiatric comorbidities
* Pharmacotherapy with psychoactive substances within the last 14 days (except treatment with SSRI/SNRIs for at least 28 days)
* Axis-I disorder according to ICD-10 and DSM 5 (except tobacco and alcohol use disorder, substance abuse with less than 2(11) criteria according to DSM-5, mild depressive episode, adaptation disorder and specific phobia within the last 12 months)
* positive urin drug screening (cannabis, amphetamine, opiates, benzodiazepines, cocaine)
* withdrawal symptoms (CIWA-R > 7)
* intoxication at time of investigation (breathalyzer > 0.3‰)
* suicidal tendency or potential danger for others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents from Mannheim/ Heidelberg who answered an open call to participate in this study
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
fMRI to assess group differences in task-specific brain activation patterns: Stress-sensitivity | fMRI measurement at one day only (day of fMRI experiment)
  Stress-sensitivity: stress task (e.g.mental rotation with and without time pressure) with social component within the MRI scanner to assess neural activation patters during the stress-task
fMRI to assess group differences in task-specific brain activation patterns: Emotion processing | fMRI measurement at one day only (day of fMRI experiment)
  Emotion-processing: emotional face-/form-matching task to assess neural activation patters of emotion processing
fMRI to assess group differences in task-specific brain activation patterns: Alcohol cue-reactivity | fMRI measurement at one day only (day of fMRI experiment)
  Alcohol cue-reactivity: pictures of alcoholic beverages to asses neural alcohol-cue reactivity

SECONDARY OUTCOMES:
Hormonal stress response using salivary cortisol level | Normal awakening response on a subject's regular week-day (0, 0.5, 8 and 14 hours after wake-up)
  Collection of saliva on a subject's regular week-day for the individual's normal cortisol awakening response and circadian rhythm (basal hypothalamic-pituitary-adrenal-function at 0, 0.5, 8 and 14 hours after wake-up).
  Cortisol awakening reaction, area under the curve and slope will therefore be calculated [nmol/L].
Hormonal stress response using salivary cortisol level | Stress response during the fMRI stress task (day of fMRI experiment, at -45, -22, -10 minutes before and 35, 45, 60, 75 and 90 minutes after onset of stress induction)
  Collection of saliva during the course of the fMRI stress task for task-induced stress effects on salivary cortisol levels (at -45, -22, -10 minutes before and 35, 45, 60, 75 and 90 minutes after onset of stress induction).
  Cortisol: Area under the curve and slope will therefore be calculated [nmol/L].
GWAS and especially glutamatergic, serotonergic single-nucleotide polymorphisms | blood sample at one day only (day of fMRI experiment)
  Genomic DNA using 40ml EDTA-blood

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Vollstaedt-Klein, Principal Investigator — CIMH Mannheim
Locations (1):
- Klinik für Abhängiges Verhalten, Zentralinstitut für Seelische Gesundheit, Mannheim, Germany

REFERENCES:
- [Derived] Gerhardt S, Berhe O, Moessnang C, Horning M, Kiefer F, Tost H, Vollstadt-Klein S. Lack of amygdala habituation to negative emotional faces in alcohol use disorder and the relation to adverse childhood experiences. Addict Biol. 2023 Jan;28(1):e13251. doi: 10.1111/adb.13251. PMID 36577733